CLINICAL TRIAL: NCT05725798
Title: Perioperative Sitagliptin Medication for Reduction of the Inflammatory Response Associated With Cardiopulmonary Bypass and Postoperative Glucose Control in Diabetic Patients Undergoing Elective Cardiac Surgery - a Pilot Study
Brief Title: Perioperative Sitagliptin Medication for Reduction of the Inflammatory Response Associated With Cardiopulmonary Bypass
Acronym: SiCa-Flam
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Sebastian Kintrup, Principal Investigator, University Hospital Muenster
Other Study IDs: 02-AnIt-19
Record Dates: First submitted 2023-01-19; First posted 2023-02-13 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: SIRS, Cardiac surgery, DPP4
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DM and Sitagliptin treatment: Cardiac surgery patients who suffer from diabetes mellitus type 2 and take Sitagliptin.
  Interventions: Drug: Sitagliptin
- DM without Sitagliptin treatment: Cardiac surgery patients who suffer from diabetes mellitus type 2 and do not take Sitagliptin.
- No DM: Cardiac surgery patients who do not suffer from diabetes mellitus type 2 and do not take Sitagliptin.

INTERVENTIONS:
Drug: Sitagliptin — Group 1 who regularly takes Sitagliptin due to diabetes mellitus type 2 continues the treatment perioperatively. Group 2 and group 3 do not take Sitagliptin.
  Groups: DM and Sitagliptin treatment

SUMMARY:
Sitagliptin is an inhibitor of the enzyme dipeptidylpeptidase-4 (DPP-4) and represents an established drug in type 2 diabetes mellitus treatment. However, Sitagliptin may also have several antiinflammatory properties. Within this study the investigators examine the effects of perioperative Sitagliptin intake on the inflammatory response after cardiopulmonary bypass.

DETAILED DESCRIPTION:
Sitagliptin is an inhibitor of the enzyme dipeptidylpeptidase-4 (DPP-4) and represents an established drug in type 2 diabetes mellitus treatment. However, Sitagliptin may also have several antiinflammatory properties. For example, it is known that DPP-4-inhibition prevents procalcitonin from being cleaved to a truncated form that lacks 2 amino acids. As the investigators described recently, truncated procalcitonin targets the CRLR-RAMP1-receptor on vascular endothelium and induces VE-cadherin-phosphorylation which leads to leakage of fluids and proteins from vessels. Furthermore, many other immunoregulatory targets such as substance p, CXCL10 or NF-kB have been reported to be modified by DPP-4. Therefore, it can be assumed that Sitagliptin possibly represents a powerful drug in inflammatory circumstances.

The aim of this study is to prove possible antiinflammatory properties by conducting an observational trial in cardiac surgery patients. All patients undergo cardiac surgery with the use of cardiopulmonary bypass (CBP) which is known to trigger a systemic inflammatory response syndrome (SIRS). Group 1 suffers from diabetes mellitus type two and regularly takes Sitagliptin which is continued perioperatively. Group 2 also suffers from diabetes mellitus type 2 but does not take Sitagliptin. Group 3 has no diabetes mellitus but also undergoes cardiac surgery. To determine the effect of Sitagliptin under inflammatory conditions deep immune phenotyping and a cytokine assay is performed from blood withdrawals 24h after surgery. Moreover, the sublingual microcirculation is measured two times after the operation.

Taking all measurements of the cellular immune system, the humoral immune system and the vasculature into account it should be possible to define the immunoregulatory effects of Sitagliptin treatment more properly.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients undergoing cardiac surgery with use of CBP and...
* Diabetes mellitus type 2 with Sitagliptin treatment or,
* Diabetes mellitus type 2 without Sitagliptin treatmet or,
* No diabetes mellitus
* Written informed consent

Exclusion Criteria:

* Diabetes mellitus type 1
* Treatment with another DPP4-inhibitor
* Treatment with GLP-1-analoga
* Emergency surgery
* Chronic or acute infection
* Pregnancy
* Participation in an interventional study trial within last 3 months
* Relationship to study investigators

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult cardiac surgery patients from University Hospital Münster who suffer from...
  * Diabetes mellitus type 2 with Sitagliptin treatment or,
  * Diabetes mellitus type 2 without Sitagliptin treatment or,
  * No diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Total norepinephrine-requirement within 24 hours after surgery | Retrospective data collection 24 hours after surgery
  Retrospective data collection from the hospital information system
Total crystalloid volume-requirement within 24 hours after surgery | Retrospective data collection 24 hours after surgery
  Retrospective data collection from the hospital information system

SECONDARY OUTCOMES:
Immune cells surface markers | Measured 24 hours after surgery
  Measured by using Cytec Aurora Flow Cytometry
Cytokine-levels | Measured 24 hours after surgery
  Measured by using multiplex immunoassay analysis.
Sublingual microcirculatory parameters: Total vessel density, Proportion of Perfused Vessels, Perfused Vessel Density, Microvascular Flow Index | Measured immediately after surgery and 24 hours after surgery
  Measured by using videomicroscopy to generate sublingual microcirculatory images.

CONTACTS AND LOCATIONS:
Overall Officials: Nana-Maria Wagner, Prof. Dr., Study Director — University Hospital Münster
Locations (1):
- University Hospital Münster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wrenger S, Kahne T, Bohuon C, Weglohner W, Ansorge S, Reinhold D. Amino-terminal truncation of procalcitonin, a marker for systemic bacterial infections, by dipeptidyl peptidase IV (DP IV). FEBS Lett. 2000 Jan 21;466(1):155-9. doi: 10.1016/s0014-5793(99)01779-2. PMID 10648832
- [Background] Brabenec L, Muller M, Hellenthal KEM, Karsten OS, Pryvalov H, Otto M, Holthenrich A, Matos ALL, Weiss R, Kintrup S, Hessler M, Dell'Aquila A, Thomas K, Nass J, Margraf A, Nottebaum AF, Rossaint J, Zarbock A, Vestweber D, Gerke V, Wagner NM. Targeting Procalcitonin Protects Vascular Barrier Integrity. Am J Respir Crit Care Med. 2022 Aug 15;206(4):488-500. doi: 10.1164/rccm.202201-0054OC. PMID 35699655
- [Background] Sablotzki A, Friedrich I, Muhling J, Dehne MG, Spillner J, Silber RE, Czeslik E. The systemic inflammatory response syndrome following cardiac surgery: different expression of proinflammatory cytokines and procalcitonin in patients with and without multiorgan dysfunctions. Perfusion. 2002 Mar;17(2):103-9. doi: 10.1177/026765910201700206. PMID 11958300
- [Derived] Hellenthal KEM, Kintrup S, Wirth T, Brabenec L, Cursiefen C, Beulen R, Hollmann K, Lehmann M, Burkard P, Roth J, Schughart K, Klotz L, Rossaint J, Meybohm P, Wagner NM. DPP4 inhibition curbs systemic inflammation. Crit Care. 2025 Aug 15;29(1):359. doi: 10.1186/s13054-025-05599-x. PMID 40817204